CLINICAL TRIAL: NCT02817555
Title: A Randomized, Controlled Trial of Costs Associated With Anemia Therapy in Hemodialysis Patients Treated With Intravenous Darbepoetin Alfa Versus Epoetin Alfa
Brief Title: Cost Comparison Study of Darbepoetin Versus Epoetin Therapy to Treat Anemia in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrea L Woodland (Other)
Responsible Party: Sponsor-Investigator, Andrea L Woodland, Clinical Pharmacist, Eastern Health, Canada
Organization: Eastern Health, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIC10.104
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: Anemia; Hemodialysis; Erythropoiesis Stimulating Agent; Cost
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Epoetin Alfa; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epoetin alfa (Active Comparator): Patients who are enrolled and randomized to the Epoetin arm will remain on their current dose and frequency. After the first hemoglobin (Hb) measurement the study algorithm will be used to guide anemia management. The subjects in this arm will remain on epoetin for the required run-in phase followed by the 12 month active phase.
  Interventions: Drug: Epoetin Alfa
- Darbepoetin alfa (Active Comparator): Patients who are enrolled and randomized to the Darbepoetin arm will have their epoetin discontinued at the end of the week preceding entry into the study and will switch to darbepoetin on the date that they would normally be receiving their next dose of epoetin.
  Switching patients to darbepoetin will be done using the conversion ratio of 200 units of epoetin to 1 μg of darbepoetin as used per week, rounded up or down to the nearest available pre-filled syringe dose available from the manufacturer.
  After the first Hb measurement the study algorithm will be used to guide anemia management. The subjects in this arm will remain on darbepoetin for the required run-in phase followed by the 12 month active phase.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Epoetin Alfa — The investigator will adjust epoetin doses as per the study algorithm during the run-in (every two weeks) and active phases (every four weeks). This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All epoetin will be administered intravenously through a hemodialysis machine port using a manufacturer-provided pre-filled syringe.
  It is not anticipated that a subject will require a dose of epoetin > 30 000 units weekly. If this occurs the dose will not be escalated any higher. Such a patient would likely meet the criteria for study withdrawal.
  Intravenous iron will be given as per the study algorithm and only one formulation of iron is used, sodium ferric gluconate.
  Other Names: Eprex
  Arms: Epoetin alfa
Drug: Darbepoetin alfa — The investigator will adjust darbepoetin doses as per the study algorithm during the run-in (every two weeks) and active phases(every four weeks). This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All darbepoetin will be administered intravenously through a hemodialysis machine port using a manufacturer-provided pre-filled syringe.
  It is not anticipated that a subject will require a dose of darbepoetin >150µg weekly. If this occurs the dose will not be escalated any higher. Such a patient would likely meet the criteria for study withdrawal.
  Intravenous iron will be given as per the study algorithm and only one formulation of iron is used, sodium ferric gluconate.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
The purpose of this study is to determine if there is a cost difference between darbepoetin alfa and epoetin alfa when used intravenously to treat anemia in hemodialysis patients.

DETAILED DESCRIPTION:
Eligible hemodialysis patients who are currently receiving an erythropoiesis stimulating agent (ESA) who enrol and sign consent will be randomized on a 1:1 basis to either remain on epoetin alfa or switch to darbepoetin alfa as their anemia therapy. Patients will be dosed with the assigned drug using a study algorithm to maintain their hemoglobin (Hb) level within the currently recommended range (100-120 g/L). There will be an initial "run in" period of a minimum of six weeks to ensure the patient's hemoglobin is stable within the target range. The trial itself will run for a subsequent twelve months (active phase). Every effort will be made to ensure that Hb stays within the target range during the study period. The primary outcome will be the total cost of each ESA therapy over the twelve month active phase. Data including Hgb, iron indices and dosing, and clinical events will be obtained from electronic sources and from the attending physicians and/or the clinical pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* age ≥19 years
* receiving in-center hemodialysis two or more times weekly
* anemia requiring erythropoiesis stimulating (ESA) agent therapy OR a hemoglobin(Hb)<100g/L in the absence of other causes of anemia
* if female, must be using an approved method of contraception or judged unable to become pregnant
* able to give informed consent

Exclusion Criteria:

* acute kidney injury likely to resolve
* plans to change to peritoneal dialysis or home hemodialysis, or planned transplant from a living donor
* expected lifespan of less than six months due to a medical condition other than chronic kidney disease
* current hematologic condition that may cause anemia
* use of medications known to cause anemia
* use of any investigational drug or androgen within 90 days of screening
* significant bleeding within 30 days of screening
* red blood cell transfusion(s) within 30 days of screening
* documented or suspected pure red cell aplasia (PRCA)
* current iron deficiency
* documented allergy or intolerance to intravenous sodium ferric gluconate
* known or probable ESA resistance
* uncontrolled hypertension
* an intention to relocate to a different dialysis center in the near future

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Woodland, BScPharm,MSc, Principal Investigator — Eastern Health, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chung EY, Palmer SC, Saglimbene VM, Craig JC, Tonelli M, Strippoli GF. Erythropoiesis-stimulating agents for anaemia in adults with chronic kidney disease: a network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 13;2(2):CD010590. doi: 10.1002/14651858.CD010590.pub3. PMID 36791280
- [Derived] Woodland AL, Murphy SW, Curtis BM, Barrett BJ. Costs Associated With Intravenous Darbepoetin Versus Epoetin Therapy in Hemodialysis Patients: A Randomized Controlled Trial. Can J Kidney Health Dis. 2017 Jun 30;4:2054358117716461. doi: 10.1177/2054358117716461. eCollection 2017. PMID 28717516

RESULTS

PARTICIPANT FLOW:
Groups:
- Epoetin Alfa: Patients who are enrolled and randomized to the Epoetin arm will remain on their pre-enrollment dose and frequency. After the first hemoglobin (Hb) measurement the study algorithm will be used to guide anemia management. The subjects in this arm will remain on epoetin for the required run-in phase followed by the 12 month active phase.
  Epoetin Alfa: The investigator will adjust epoetin doses as per the study algorithm during the run-in (every two weeks) and active phases (every four weeks). This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All epoetin will be administered intravenously through a hemodialysis machine port using a manufacturer-provided pre-filled syringe.
  It is not anticipated that a subject will require a dose of epoetin > 30 000 units weekly. If this occurs the dose will not be escalated any higher. Such a patient would likely meet the criteria for study withdrawal.
- Darbepoetin Alfa: Patients who are enrolled and randomized to the Darbepoetin arm will have their epoetin discontinued at the end of the week preceding entry into the study and will switch to darbepoetin on the date that they would normally be receiving their next dose of epoetin.
  Switching patients to darbepoetin will be done using the conversion ratio of 200 units of epoetin to 1 μg of darbepoetin as used per week, rounded up or down to the nearest available pre-filled syringe dose available from the manufacturer.
  After the first Hb measurement the study algorithm will be used to guide anemia management. The subjects in this arm will remain on darbepoetin for the required run-in phase followed by the 12 month active phase.
  Darbepoetin alfa: The investigator will adjust darbepoetin doses as per the study algorithm during the run-in (every two weeks) and active phases(every four weeks). This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
Period: Overall Study
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Started | 24 | 26
Completed | 21 | 21
Not Completed | 3 | 5
Not completed — Death | 1 | 3
Not completed — moved away | 1 | 0
Not completed — transplant | 1 | 1
Not completed — changed to Peritoneal Dialysis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Epoetin Alfa: Patients who are enrolled and randomized to the Epoetin arm will remain on their current dose and frequency. After the first hemoglobin (Hb) measurement the study algorithm will be used. The subjects will remain on epoetin for the required run-in phase followed by the 12 month active phase.
  The investigator will adjust epoetin doses as per the study algorithm during the run-in and active phases. This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All epoetin will be administered intravenously through a hemodialysis machine port using a manufacturer-provided pre-filled syringe.
  It is not anticipated that a subject will require a dose of epoetin > 30 000 units weekly. If this occurs the dose will not be escalated any higher.
  Intravenous iron will be given as per the study algorithm and only one formulation of iron is used, sodium ferric gluconate.
- Darbepoetin Alfa: Patients who are randomized to the Darbepoetin arm will have their epoetin and will switch to darbepoetin on the date that they would normally be receiving their next dose of epoetin.
  Switching patients will be done using the conversion ratio of 200 units of epoetin to 1 μg of darbepoetin as used per week, rounded to the nearest pre-filled syringe available from the manufacturer.
  After the first Hb measurement the study algorithm will be used.
  The investigator will adjust darbepoetin doses as per the study algorithm during the run-in and active phases. This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All darbepoetin will be administered intravenously through a hemodialysis machine port.
  It is not anticipated that a subject will require a dose of darbepoetin >150µg weekly. If this occurs the dose will not be escalated any higher.
  Intravenous iron will be given as per the study algorithm, sodium ferric gluconate.
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa | Darbepoetin Alfa | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (13.3) | 61 (15.1) | 60.49 (13.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 11 | 20 | 31
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 26 | 50

OUTCOME MEASURES:

1. Primary Outcome: Cost of Erythropoiesis Stimulating Agent
Description: total cost over 12 months in Canadian dollars
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: dollars Canadian
Groups:
- Epoetin Alfa: Patients who are enrolled and randomized to the Epoetin arm will remain on their current dose and frequency. After the first hemoglobin (Hb) measurement the study algorithm will be used to guide anemia management. The subjects in this arm will remain on epoetin for the required run-in phase followed by the 12 month active phase.
  Epoetin Alfa: The investigator will adjust epoetin doses as per the study algorithm during the run-in (every two weeks) and active phases (every four weeks). This will continue until the 12 month active phase is complete or the patient is withdrawn from the study.
  All epoetin will be administered intravenously through a hemodialysis machine port using a manufacturer-provided pre-filled syringe.
  It is not anticipated that a subject will require a dose of epoetin > 30 000 units weekly. If this occurs the dose will not be escalated any higher. Such a patient would likely meet the criteria for study withdrawal.
  Intravenous iron will be given as per the
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
dollars Canadian | 4178.70 [2416.37 to 5955.12] | 2302.92 [1177.86 to 4218.93]

2. Secondary Outcome: Hemoglobin
Description: median hemoglobin (g/L) over 12 months
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
g/L | 108 [106 to 112.7] | 109.8 [105.9 to 116.1]

3. Secondary Outcome: Ferritin
Description: mean ferritin (ug/L) over 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
ug/L | 847.58 (272.88) | 726.29 (377.13)

4. Secondary Outcome: Transferrin Saturation (TSAT)
Description: median TSAT (%) over 12 months
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: percentage saturation
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
percentage saturation | 26.71 [22.46 to 32.33] | 28.58 [23.9 to 33.75]

5. Secondary Outcome: Iron Dose
Description: median weekly iron dose (mg) over 12 months
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: mg/week
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
mg/week | 40.36 [20.83 to 59.9] | 41.67 [19.53 to 70.96]

6. Secondary Outcome: Iron Cost
Description: total iron cost over 12 months in Canadian dollars
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: canadian dollars
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 26
canadian dollars | 726.56 [375 to 1078.13] | 750 [351.56 to 1277.34]

ADVERSE EVENTS:
Time Frame: Run in phase and 12 month study period.
Arm/Group | Epoetin Alfa | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 1/24 | 3/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 0/24 | 0/26

LIMITATIONS AND CAVEATS:
Did not recruit planned number, incomplete follow up in 8 subjects, cannot be generalized to centres without pre-defined dosing algorithms, non-dialysis CKD, or sc administration of ESAs. Trial looked at drug acquisition cost only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No